CLINICAL TRIAL: NCT07293091
Title: A Randomized, Double-Blind, Crossover Study to Assess the Appearance of Amino Acids in Circulation Following Acute Consumption of Two Protein Beverages
Brief Title: Assessing the Appearance of Amino Acids in Circulation Following Consumption of Protein Beverages
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2528
Record Dates: First submitted 2025-12-02; First posted 2025-12-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Tolerability; Appetite; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - Protein Beverage (Experimental): Protein powder mixed into 8 oz of water
  Interventions: Dietary Supplement: Protein Powder
- Active Control - Protein Beverage (Active Comparator): Control protein powder mixed into 8 oz of water
  Interventions: Dietary Supplement: Control Protein Powder

INTERVENTIONS:
Dietary Supplement: Protein Powder — Contains 30 g of protein
  Arms: Experimental - Protein Beverage
Dietary Supplement: Control Protein Powder — Contains 30 g of protein
  Arms: Active Control - Protein Beverage

SUMMARY:
The objective of this study is to compare the appearance of amino acids in circulation following consumption of two protein beverages in adults. Secondary objectives of this study are to assess changes in gastrointestinal tolerability, glycemia, markers of subjective and physiological appetite, and nausea.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, between 25 and 54 years of age.
* 2. Individual has a body mass index (BMI) of 22.5 to 32.5 kg/m2. Only 5 participants will have a BMI of 30 to 32.5 kg/m2.
* 3. Individual is judged by the Investigator to be in generally good health on the basis of medical history and screening measurements.
* 4. Individual is willing and able to undergo the scheduled study procedures.
* 5. Individual is willing to maintain usual physical activity level for the duration of the study and not to engage in vigorous physical activity for at least 24 hours prior to each clinic visit.
* 6. Individual is willing to abstain from alcohol consumption for at least 24 hours prior to each clinic visit.
* 7. Individual understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* 1. Individual has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
* 2. Individual has poor venous access and is not a good candidate for serial blood draws.
* 3. Use of tobacco/nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 6 months of visit 1.
* 4. Individual has anemia (hemoglobin <9 g/dL for females and <11 g/dL for males).
* 5. Individual has a clinically significant medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results. Health conditions may include history or presence of clinically important gastrointestinal, cardiac, renal, hepatic, endocrine (e.g., type 1 or type 2 diabetes mellitus), pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
* 6. Individual had a recent (within two weeks of screening) episode of acute gastrointestinal illness such as nausea, vomiting, or diarrhea.
* 7. Individual has a history of frequent diarrhea or constipation that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
* 8. Individual has a history of stomach or gastrointestinal surgery (e.g., gastric bypass, cholecystectomy) that in the opinion of the Investigator, could interfere with evaluation of the study outcomes.
* 9. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
* 10. Individual uses medications (over-the counter or prescription) or dietary supplements known to influence gastrointestinal motility or digestion including laxatives, enemas, or suppositories; digestive enzyme supplements, proton pump inhibitors, H2 blockers, alpha-glucosidase inhibitors, antacids; prokinetic drugs; anti-diarrheal agents, anti-cholinergic drugs including anti-spasmodics; and fiber supplements. A 14-day washout phase prior to visit 2 (day 0) is allowed for participants taking any of these products.
* 11. Unstable use (initiation or change in dose) within 30 days of visit 1 of sex hormones. Multiphasic hormonal contraceptives in which the amount of sex hormone in the active pill varies by week (i.e., biphasic, triphasic, quadriphasic) are considered unstable doses of sex hormones and are exclusionary.
* 12. Use of any weight loss medication (including over-the-counter medications and/or supplements) within 30 days of visit 1.
* 13. Individual has used an alpha-blocker, beta-blocker, or high-dose diuretic within 30 days of visit 1. Unstable use (initiation or change in dose) within 30 days of visit 1 of other antihypertensive medications is also exclusionary.
* 14. Unstable use (initiation or change in dose) within 90 days of visit 1 of thyroid hormone replacement medications.
* 15. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg).
* 16. Individual has a recent history of cancer in the prior 2 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
* 17. Individual has signs or symptoms of an active infection of clinical significance or has taken antibiotics within 5 days prior to any visit (washout is permitted for re-scheduling of the clinic visit).
* 18. Individual regularly consumes (≥2 servings per week) protein supplements (including collagen) within 2 weeks of visit 2.
* 19. Individual has extreme dietary habits (e.g., ketogenic, very high protein, very high fiber, vegan, vegetarian).
* 20. Individual is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* 21. Individual has a known allergy or sensitivity to any ingredients in the study beverages or meals.
* 22. Individual has been exposed to any non-registered drug product within 30 days of the first screening visit.
* 23. Individual has a current or recent history (past 12 months of screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
* 24. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 25 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Total Amino Acid net incremental area under the curve (niAUC) | 5-12 hours post-beverage consumption
  Difference between conditions in the niAUC for the total amino acid level in plasma

SECONDARY OUTCOMES:
Total Amino Acids area under the curve (AUC) | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in AUC for the total amino acid level in plasma
Total Amino Acids niAUC | 0-5 hours and 0-12 hours
  Difference between conditions in the niAUC for the total amino acid level in plasma
Maximum concentration for total amino acids | 0-12 hours
  Difference between conditions in the maximum concentration for total amino acids in plasma
Baseline-adjusted maximum concentration for total amino acids | 0-12 hours
  Difference between conditions in the baseline-adjusted maximum concentration for total amino acids in plasma
Time to maximum concentration for total amino acids | 0-12 hours
  Differences between conditions in the time to maximum concentration for total amino acid levels in plasma
Glucagon-like peptide-1 AUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the AUC for glucagon-like peptide-1
Glucagon-like peptide-1 niAUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the niAUC for glucagon-like peptide-1
Peptide YY AUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the AUC for peptide YY
Peptide YY niAUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the niAUC for peptide YY
Ghrelin AUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the AUC for ghrelin
Ghrelin niAUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the niAUC for ghrelin
Glucose-dependent insulinotropic polypeptide AUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the AUC for glucose-dependent insulinotropic polypeptide
Glucose-dependent insulinotropic polypeptide niAUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Differences between conditions in the niAUC for glucose-dependent insulinotropic polypeptide
Markers of subjective appetite AUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Difference between conditions in the AUC for markers of subjective appetite (hunger, fullness, desire to eat, and prospective consumption) measured by the visual analog scale
Markers of subjective appetite niAUC | 0-5 hours, 5-12 hours, and 0-12 hours
  Difference between conditions in the niAUC for markers of subjective appetite (hunger, fullness, desire to eat, and prospective consumption) measured by the visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ocean Wellness Center, Miami Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided